CLINICAL TRIAL: NCT02213302
Title: Effects of Premedication by Midazolam on Preoperative Anxiety for Emergency Surgery
Brief Title: Premedication by Midazolam for Emergency Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-000873-38; PROM 2012_30 (Other: University hospital, Lille)
Record Dates: First submitted 2014-07-02; First posted 2014-08-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Anxiety
Keywords: premedication; preoperative anxiety; salivary cortisol level; anxiety visual analog scale
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isotonic serum (Placebo Comparator): placebo administration
  Interventions: Drug: placebo administration; Drug: midazolam intravenous administration
- Midazolam (Active Comparator): midazolam intravenous administration 0.02mg/kg
  Interventions: Drug: placebo administration; Drug: midazolam intravenous administration

INTERVENTIONS:
Drug: placebo administration
  Other Names: isotonic saline serum intravenous administration
Drug: midazolam intravenous administration
  Other Names: hypnovel

SUMMARY:
Preoperative anxiety is a subjective and painful experience and may have adverse psychological consequences and complicate anesthetic management. The aim of the study is to show the effect of premedication by midazolam on preoperative anxiety assessed by a visual analog scale and by measuring salivary cortisol levels. This study was a monocentric, prospective, blind randomized placebo controlled clinical study. Sixty patients, aged 18 to 79 years, to undergo elective surgery under general anesthesia with tracheal intubation must be enrolled and randomized to receive midazolam (0.02mg/kg) or placebo. The primary outcome is the reduction in anxiety assessed by a visual analog scale. The secondary outcomes are the reduction in salivary cortisol levels, the overall level of anxiety and the evaluation of respiratory and hemodynamic adverse effects of midazolam.

ELIGIBILITY:
Inclusion Criteria:

* major patient undergoing elective surgery under general anesthesia with tracheal intubation
* Anesthesia state 1 and 2
* preoperative fasting for 6 hours
* information and signed consent
* social security
* non pregnant women

Exclusion Criteria:

* anesthesia state above 3
* midazolam sensibility
* pregnant or breastfeeding women
* ICU patients
* no consent
* pediatric surgery
* no social security
* no tracheal intubation
* required premedication in placebo group or midazolam sensibility in premedication group

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale of anxiety | baseline, up to the end of support in recovery room
  visual scale rated from 0 to 10 to describe the intensity of anxiety simple and reproducible measurement for a short period

SECONDARY OUTCOMES:
salivary cortisol level | baseline and at the entrance in operating room
  biologic measurement non-invasive, inexpensive and easy to perform. two determinations before and after premedication (at least 20 minutes)
Global anxiety | baseline
  rated from 4 to 20 for global anxiety and from 2 to 10 for information request anxiety is high above 10 for women and 12 for men
Patient's satisfaction | at the end of the support in recovery room
  rated from 1 for bad management to 5 for excellent management assessed at the output of the recovery room
Intraoperative consumption of hypnotics and opioids | at anesthesia induction up to 10 minutes
  Cumulative dose of hypnotics and opioids reduced to dose per kilogram
Comfort induction | at anesthesia induction
  rated from 1 for deep discomfort to 5 for good comfort
Intubation score | after intubation
  Rated from 1 bed conditions for intubation to 5 for excellent conditions
Adverse midazolam effects | baseline up to the end of support in recovery room
  assessed by variations of arterial pressure, heart rate, respiratory rate, oxygen saturation and end tidal of carbon dioxide for hemodynamics and respiratory adverse effects assessed by Observer's assessment of alertness/sedation for deep of sedation rated from 1 sleeping patient to 5 for awake patient
Output score of recovery room (Aldrete score) | at the end of support in recovery room
  rated from 0 to 10 essential for the output of recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Elise Blondé-Zoonekynd, Physician, Principal Investigator — University Hospital, Lille
Locations (1):
- Emergency, University Hopital, Lille, France

REFERENCES:
- [Result] Sun GC, Hsu MC, Chia YY, Chen PY, Shaw FZ. Effects of age and gender on intravenous midazolam premedication: a randomized double-blind study. Br J Anaesth. 2008 Nov;101(5):632-9. doi: 10.1093/bja/aen251. Epub 2008 Sep 4. PMID 18772216
- [Result] Vogelsang J. The Visual Analog Scale: an accurate and sensitive method for self-reporting preoperative anxiety. J Post Anesth Nurs. 1988 Aug;3(4):235-9. No abstract available. PMID 2457102
- [Result] Bauer KP, Dom PM, Ramirez AM, O'Flaherty JE. Preoperative intravenous midazolam: benefits beyond anxiolysis. J Clin Anesth. 2004 May;16(3):177-83. doi: 10.1016/j.jclinane.2003.07.003. PMID 15217656
- [Result] Jerjes W, Jerjes WK, Swinson B, Kumar S, Leeson R, Wood PJ, Kattan M, Hopper C. Midazolam in the reduction of surgical stress: a randomized clinical trial. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Nov;100(5):564-70. doi: 10.1016/j.tripleo.2005.02.087. PMID 16243241
- [Result] Wattier JM, Barreau O, Devos P, Prevost S, Vallet B, Lebuffe G. [Measure of preoperative anxiety and need for information with six issues]. Ann Fr Anesth Reanim. 2011 Jul-Aug;30(7-8):533-7. doi: 10.1016/j.annfar.2011.03.010. Epub 2011 May 23. French. PMID 21602018
- [Result] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Result] Reves JG, Fragen RJ, Vinik HR, Greenblatt DJ. Midazolam: pharmacology and uses. Anesthesiology. 1985 Mar;62(3):310-24. PMID 3156545
- [Result] Zalunardo MP, Ivleva-Sauerborn A, Seifert B, Spahn DR. [Quality of premedication and patient satisfaction after premedication with midazolam, clonidine or placebo : Randomized double-blind study with age-adjusted dosage]. Anaesthesist. 2010 May;59(5):410-8. doi: 10.1007/s00101-010-1695-9. German. PMID 20224951